CLINICAL TRIAL: NCT02734784
Title: Clinical and Microbiological of Antimicrobial Photodynamic Therapy on Surgical Treatment of Chronic Periodontitis: a Double-blind Split-mouth Randomized Controlled Clinical Trial.
Brief Title: Treatment of Chronic Periodontitis With Repeated Adjunctive Antimicrobial Photodynamic Therapy
Acronym: TCPWRAAPT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Sergio Luis Scombatti de Souza, Dr., University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 14/09801-9
Record Dates: First submitted 2016-04-06; First posted 2016-04-12 (Estimated); Last update posted 2016-04-12 (Estimated); Status verified 2016-04

CONDITIONS: Chronic Periodontitis
MeSH Terms: conditions — Chronic Periodontitis | interventions — Photochemotherapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Photodynamic Therapy and SRP (Experimental)
  Interventions: Procedure: Photodynamic Therapy
- SRP and Sham Photodynamic Therapy (Sham Comparator)
  Interventions: Procedure: Sham Photodynamic Therapy

INTERVENTIONS:
Procedure: Photodynamic Therapy — After a surgical access, the periodontal pockets of teeth selected to receive antimicrobial photodynamic therapy (aPDT) will be irrigated with distilled water. Shortly thereafter, the dye will be applied (phenothiazine hydrochloride- 10mg/mL) from the bottom of the pocket. After 1 minute, irrigation will be performed with distilled water to remove the excess of dye. The stained area will be irradiated with a diode laser (660 nm and a 60 mW/cm²). Six sites per tooth under treatment will be irradiated (10 seconds/ site). Teeth with furcation lesion will increase over 60 seconds into the lesion. Before the application, the supragingival plaque will be removed.
  Arms: Photodynamic Therapy and SRP
Procedure: Sham Photodynamic Therapy — After a surgical access, the periodontal pockets of teeth selected will receive a simulation of antimicrobial photodynamic therapy (aPDT): irrigation with distilled water and simulated laser application. Before the application, the supragingival plaque will be removed.
  Arms: SRP and Sham Photodynamic Therapy

SUMMARY:
Chronic periodontitis (CP) is an infectious disease resulting in inflammation of the supporting structures of the teeth, progressive loss of bone loss and insertion. The aim of this study is to evaluate the effects of antimicrobial Photodynamic Therapy (aPDT) as adjuvant to periodontal surgery treatment (PST) in patients diagnosed with generalized severe chronic periodontitis (GSCP). Twenty patients with a clinical diagnosis of CP will be treated in a split-mouth design study to either aPDT associated with surgical access for scaling and root planning (SASRP) or SASRP only. aPDT will be performed by using a laser light source with 690 nm wavelength associated with a phenothiazine photosensitizer. The applications will occur in only one episodes. All patients will be monitored for 30 and 90 days after PST. Clinical assessment of plaque index, probing depth, clinical attachment level and bleeding on probing will be performed at baseline (pre-intervention period) and 30 and 90 days after the PST. Subgingival plaque samples will be collected (at baseline and 30 and 90 days after the PST) and the counts of 40 subgingival species will be determined using DNA-DNA checkerboard hybridization. Data obtained will be statistically analyzed.

DETAILED DESCRIPTION:
Non-Surgical Periodontal Therapy

Seven days prior to the non-surgical periodontal therapy, periapical radiographs will be taken from the whole mouth of all patients. They will be set in an oral hygiene program (OHP) according to their specific needs. In this program, patients will be instructed about an effective self-performed plaque control, including information about the Bass Technique (Bass, 1954) and interproximal cleaning with dental floss and interdental brushes. They will be also motivated to brush the dorsal surface of the tongue once a day and will receive a dentifrice that shall be used throughout the experimental period (Colgate Total®, Anakol Ind. Com Ltda - Brazil's Kolynos - Colgate Palmolive Co., Sao Bernardo do Campo, SP, Brazil). After the OHP, subjects will undergo the assessment of clinical periodontal parameters previously described and the collection of subgingival plaque and GCF in selected sites (baseline) will be performed. Shortly, patients will receive supragingival scaling and coronal polishing with prophy cup on all the teeth present in the oral cavity. The non-surgical periodontal therapy will initiate 7 days after the OHP and initial supragingival scaling. Within 24 hours, a specialist in Periodontics will perform supra and subgingival scaling and root planing of all teeth with periodontal involvement, using hand (Gracey Curettes, Hu-Friedy, Chicago, IL, USA) and ultrasonic instruments. The instrumentation will be performed on each quadrant until achievement of an adequate cleaning and root planing, which will be verified with a dental explorer. Individuals will receive professional prophylaxis biweekly during three months after the end of the nonsurgical periodontal therapy. On biweekly follow-up visits, patient's cooperation will be monitored by verifying the status of oral hygiene.

Surgical Periodontal Therapy

The flap operations are performed 8 weeks after the start of the basic preparation. Patients will be monitored clinically and sites that present PS ≥ 5mm and SS presence will undergo surgical therapy scraping retail. Surgical procedures will be performed by a specialist in Periodontics. Initially patients will be subjected to extra-oral antisepsis with chlorhexidine 2% and intraoral through mouthwash with chlorhexidine 0.12%. The region to be operated infiltrative receive local anesthesia with lidocaine 2% solution, and 1: 100,000 epinephrine. The following will be performed intra-sulcular incision with a scalpel blade at 15C covering the site with PS ≥ 5mm and the adjacent teeth. A mucoperiosteal flap will be performed until the exposure of the bone crest and subgingival deposits of calculation and / or granulation tissue are removed by conventional Gracey curettes with RAR and Mini Five, numbers 5/6, 7/8, and 11/12 13/14 (Hu-Friedy, Chicago, IL, USA) and ultrasonic devices. Shortly after completion of the RAR starts to tfdA the operated region in the selected adjuvant therapy for this group. Completed therapy, the flap will be positioned in the same place of origin and stabilized with simple sutures through wire Vicryl 5-0. In order to avoid painful symptoms will be prescribed analgesics (Paracetamol 750mg, 01 tablet every 6 hours for 48 hours). They will also be prescribed soft oral rinses with 0.12% chlorhexidine digluconate, 2 times a day for 14 days. The sutures are removed after 7 days. Being performed weekly supragingival plaque control in the first month and monthly until completing 3 after surgical intervention months.

Antimicrobial photodynamic Therapy

After surgical access and realization of flap RARÎ, surgical sites selected to receive the TfdA will be irrigated with saline will be dried with sterile gauze, a period of 10 minutes and waited, until there is no more bleeding. Soon after, will be applied fotossintentizador hydrochloride phenothiazine, whose main component is the toluidine blue at a concentration of 10mg / mL (Helbo Blue, Helbo Photodynamic Sytems, Grieskirchen, Austria), which will be in contact for 3 minutes. Posteriorly, irrigation will be performed with saline solution for removal of the excess fotossensitizador and colored areas are irradiated with a laser diode of wavelength 660 nm, maximum power 60 mW / cm2 and an energy density of 0,6J / cm2 ( Helbo therapielaser, Helbo Photodynamic Systems GmbH & Co KG, Grieskirchen, Austria), for 60 seconds per site. The treatment is carried out in 6 sites on the teeth, totaling six minutes of application of laser light per tooth. Teeth with furcation lesion will increase more 60 seconds into the lesion.

Each patient will be impressed with alginate in order to obtain models of the dental arches and elaborate a guide plate made of acetate. This plate will present grooves that will be used as references to standardize the insertion and tilt of the automated periodontal probe (Florida Probe System, Florida Probe Corporation, Gainesville, FL, USA). The visible plaque index for each patient, rated dichotomously (O'Leary et al. 1972), will be determined by the percentage of tooth surfaces with deposits of plaque stained with disclosing solution.

Clinical monitoring

The following clinical periodontal parameters will be assessed at 6 sites of each tooth (mesio-buccal, buccal, disto-buccal, mesio-lingual, lingual and disto-lingual): (i) probing pocket depth (PPD): it will be measured from the gingival margin to the bottom of the pocket; (ii) gingival recession (GR): it will be measured from the enamelcement junction to the bottom of the pocket; (iii) clinical attachment level (CAL): it will be measured as PPD + GR (GR will be equal to 0 whenever the cementenamel junction is covered); (iv) bleeding on probing (BOP): it will be evaluated dichotomously: the presence of the bleeding will be considered positive when occurring within 30 seconds from the insertion of the probe for probing depth; (v) Plaque index (PI): it will be evaluated dichotomously. BOP, PPD, CAL and GR will be measured at six sites per tooth (mesio-buccal, buccal, disto-buccal, disto-lingual, lingual and mesio-lingual). All probing measurements will be performed using an automated periodontal probe.

The clinical periodontal parameters and the plaque index of each patient will be recorded at baseline (pre-intervention), as well as +30 and +90 days after the non-surgical periodontal therapy. The Kappa index will be used to evaluate the examiner calibration on clinical periodontal parameters collection in order to calculate the intra-examiner agreement. According to the World Health Organization (WHO) criteria for diagnosis, the acceptable Kappa index of agreement must be greater than or equal to 0.85 (WHO, 1997). This level of agreement will be used for calibration of the examiner in this project. Ten patients, each one showing at least two pairs of contralateral single-rooted teeth with PD ≥ 5 mm on interproximal sites, will be selected to calibrate the examiner. Each patient will be evaluated on two separate occasions 48 hours apart in order to obtain the intra-examiner reliability through the Kappa index.

Microbiological monitoring

At baseline and +30 and +90 days after the non-surgical periodontal therapy, samples of subgingival plaque will be obtained from eight interproximal sites of each patient. Samples will be individually analyzed for their content of 40 subgingival bacterial species using the checkerboard DNA-DNA hybridization technique (Socransky et al., 2004a; Socransky et al., 2004b). The selected teeth will be isolated with sterile cotton rolls and dried with air jets. Then, the supragingival plaque will be carefully removed using a sterile curette. Another sterile curette will be used to collect the subgingival plaque, starting from the bottom of the periodontal pocket to its coronal portion. The samples will be stored in sterilized Eppendorf tubes and will be processed at the Microbiology Laboratory of the Guarulhos University (UNG, Guarulhos, SP, Brazil).

Statistical analysis

The normality and homoscedasticity of the data obtained will be checked. Comparisons within groups and among groups at different time intervals will be performed through parametric or non-parametric appropriate tests. The significance level will be set at 5% in all tests. All calculations will be performed by SPSS software (SPSS, Chicago IL, USA).

ELIGIBILITY:
Inclusion Criteria:

* Subjects with >35 years old
* A minimum of 15 teeth present
* One pair of posterior teeth in opposite sides with proximal sites showing probing depth and clinical attachment level ≥ 5 mm.

Exclusion Criteria:

* Positive history of antibiotic-therapy in the last six months
* Positive history of basic periodontal treatment in the last six months
* Systemic disease that can interfere with the progression of disease or response to treatment (eg, diabetes, immune disorders)
* Extensive prosthetic involvement
* Need for antibiotic prophylaxis for performing routine dental procedures
* Use of anti-inflammatory drugs for long periods of time
* Smoking
* Pregnancy

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-02; Primary Completion 2015-11 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in clinical attachment level at +120 days | The clinical periodontal parameter will be recorded at baseline (pre-intervention) and +120 days after the surgical periodontal therapy.

SECONDARY OUTCOMES:
Change from baseline in counts of 40 subgingival bacterial species at +30 and +120 days | Microbiological monitoring (at baseline and +30 and +120 days after the surgical periodontal therapy) using the checkerboard DNA-DNA hybridization
Numbers of patients requiring additional periodontal treatment at +120 days. | Considering each group separately, it will be evaluate the number of patients presenting at least a site with PPD≥5 mm and positiveBOP at 120 days post-therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Sérgio S. de Souza, Dr., Principal Investigator — University of Sao Paulo

REFERENCES:
- [Derived] Martins SHL, Novaes AB Jr, Taba M Jr, Palioto DB, Messora MR, Reino DM, Souza SLS. Effect of surgical periodontal treatment associated to antimicrobial photodynamic therapy on chronic periodontitis: A randomized controlled clinical trial. J Clin Periodontol. 2017 Jul;44(7):717-728. doi: 10.1111/jcpe.12744. Epub 2017 Jun 29. PMID 28498507